CLINICAL TRIAL: NCT02888249
Title: Behavioral Economic Purchasing Decisions for Cigarettes of Varied Compositions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00107178; 5R01DA042527 (NIH)
Record Dates: First submitted 2016-08-23; First posted 2016-09-02 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2021-01

CONDITIONS: Tobacco Use Disorder; Substance-Related Disorders
Keywords: Tobacco withdrawal; Autonomic Agents
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cigarette W (Experimental): Altered composition cigarettes
  moisture = 12.20 %, tar = 10.40 mg/cigarette, total particulate matter = 12.0 mg/cigarette, high sugar content
  Interventions: Other: Altered composition cigarette
- Cigarette X (Experimental): Altered composition cigarettes
  moisture = 12.10 %, tar = 8.60 mg/cigarette, total particulate matter = 9.60 mg/cigarette, low sugar content
  Interventions: Other: Altered composition cigarette
- Cigarette Y (Experimental): Altered composition cigarettes
  moisture = 13.20 %, tar = 9.10 mg/cigarette, total particulate matter = 10.10 mg/cigarette, low sugar content
  Interventions: Other: Altered composition cigarette
- Cigarette Z (Experimental): Altered composition cigarettes
  moisture = 13.60 %, tar = 8.10 mg/cigarette, total particulate matter = 9.10 mg/cigarette, low sugar content
  Interventions: Other: Altered composition cigarette

INTERVENTIONS:
Other: Altered composition cigarette — This double-blind study will systematically determine the abuse liability of altered composition cigarettes using a behavioral economics abuse-liability approach. Altered composition cigarettes (e.g., cigarettes differing in casings, sugars, tar levels, moisture) may result in decreased intake and decreased dependence, although critical questions remain regarding the abuse-liability of altered composition cigarettes, whether exposure to these cigarettes reduces use, and whether altered composition cigarettes will substitute for standard cigarettes. The addictive effects and abuse liability of altered composition cigarettes, therefore, are not well understood, and will be tested in this study.

SUMMARY:
The purpose of this study is to determine whether the abuse liability of cigarettes with altered composition (cigarettes differing in composition; e.g., tar levels, amount of sugar, casings) is reduced relative to standard composition cigarettes.

DETAILED DESCRIPTION:
The proposed study will determine the abuse liability of altered composition cigarettes compared to standard cigarettes using a behavioral economics abuse-liability approach. Behavioral economic demand analysis constitutes a comprehensive examination of drug reinforcement and abuse liability. Laboratory determination of cigarette consumption under various response requirements will occur before and after 3 weeks of at-home exposure, with participants randomized to cigarettes varying in composition to determine the role of experience on the abuse-liability of various cigarettes. Abuse liability will be assessed by 2 essential demand metrics: lower demand intensity and increased demand elasticity, as well as other demand metrics and subjective ratings of "liking". The study will also determine the degree to which altered composition cigarettes may substitute for standard composition cigarettes - testing whether an altered composition policy would achieve the goal of reducing standard cigarette consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Smoke at least five cigarettes per day
3. Have an expired carbon monoxide level of more than 8 ppm or a urinary cotinine level of more than 100 ng per milliliter
4. Have a Fagerström Test for Nicotine Dependence score of at least 5 upon screening

Exclusion Criteria:

1. The intention to quit smoking in the next 30 days
2. The use of other tobacco products in addition to machine-manufactured cigarettes on more than 9 of the previous 30 days
3. Use of "roll your own" cigarettes as an exclusive form of smoking
4. A serious medical or psychiatric disorder or unstable condition
5. Any positive toxicological screening for illicit drugs other than cannabis will be excluded
6. Women who are pregnant, plan to become pregnant or are breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Demand Intensity: Number of cigarette puffs obtained at the lowest fixed ratio value | 3 weeks after initiation of home exposure period
  The primary behavioral economic demand curve metric (demand intensity, i.e., number of cigarette puffs obtained at the lowest fixed ratio value assessed) derived from cigarette consumption in the laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Johnson, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Bayview Campus, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No